CLINICAL TRIAL: NCT06841250
Title: Early Changes in OCT Biomarkers After the First Intravitreal Anti-VEGF Injection in Treatment-naïve DME
Status: Enrolling by invitation | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nada Essam Ahmed, Nada Essam Ahmed, Sohag University
Other Study IDs: Soh-Med--25-1-08MS
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Early OCT Biomarker Changes in Response to Anti-VEGF

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- DME patients who are treatment-naïve: The collected OCT data will include the following biomarkers:
  * Determining the type of DME (diffuse, cystoid, serous retinal detachment).
  * Mean central subfield thickness (CST).
  * Presence, location and height of macular Intraretinal cystoid spaces (ICS).
  * Presence of Subfoveal neuroretinal detachment (SND) and height of serous macular detachment.
  * The presence and size, and localization of hyperreflective foci (HF) within the retina.
  * The disorganisation of the inner retinal layers (DRIL).
  * The presence of vitreomacular traction.
  * The integrity of the outer retinal layers, (ellipsoid zone (EZ) and external limiting membrane (ELM)).
  Interventions: Procedure: intravitreal injection of anti-VEGF

INTERVENTIONS:
Procedure: intravitreal injection of anti-VEGF — Ranibizumab is injected into the vitreous under aseptic conditions as part of routine DME treatment

SUMMARY:
A retrospective, observational, hospital-based study which will be conducted in the Department of Ophthalmology, Sohag University Hospital, Egypt.

DETAILED DESCRIPTION:
Aim of the work To evaluate early changes in OCT biomarkers and visual acuity in treatment-naïve patients with diabetic macular oedema after the first intravitreal antiVEGF injection.

Patients and methods Study Design A retrospective, observational, hospital-based study which will be conducted in the Department of Ophthalmology, Sohag University Hospital, Egypt.

Patients This study will include 50 eyes with center-involving DME (CI-DME) of patients who received their 1st AntiVEGF injection as a routine treatment in the Department of Ophthalmology, Sohag University Hospital.

Inclusion Criteria

1. Diabetic patients with center-involving DME (CI-DME) who are treatment-naïve.
2. Central macular thickness (CMT) of 300 microns or more will be accepted as CI-DME.

Exclusion Criteria

1. Media opacities affecting OCT imaging (corneal pathologies, dense cataracts, vitreous opacities, etc).
2. Patients with any other retinal vascular diseases (retinal vein occlusion, central serrous chorioretinopathy, age-related macular degeneration, etc).
3. Patients who have had previous intravitreal injections or Laser treatment.
4. Patients who underwent previous vitreoretinal surgeries.
5. Patients with recent history of undergoing cataract surgery.
6. Patients with uncontrolled glaucoma or ocular inflammations (eg: vitritis). 4

Methods

We will analyze the medical records of the study participants before and after injection and the collected data will include:

A. History:

Patient age, gender, duration and treatment of diabetes mellitus, visual impairment history, ocular/systemic comorbidities, topical/systemic drug intake, previous ocular/systemic interventional procedures or surgery.

B. Medical Examination and Laboratory investigations:

Blood Pressure, Lipid profile, HbA1c will be measured.

C. Full ophthalmological examination:

Data recorded from the preoperative ophthalmic examination of the studied eye, which includes:

1. Best corrected visual acuity (BCVA): Snellen visual acuities will be presented as Snellen decimal notation.
2. Intraocular pressure (IOP) measured by I-Care rebound tonometer.
3. Slit lamp examination of the anterior segment and angle of the anterior chamber.
4. Fundus examination by indirect ophthalmoscope and slit lamp biomicroscopy with documentation of the stage of diabetic retinopathy.

D. OCT imaging:

OCT images and data will be collected and analysed from the electronic medical reports for all patients at 3 points:

1. Before injection (within one week before the procedure).
2. Two weeks after injection.
3. One month after injection. 5

The collected OCT data will include the following biomarkers:

* Determining the type of DME (diffuse, cystoid, serous retinal detachment).
* Mean central subfield thickness (CST).
* Presence, location and height of macular Intraretinal cystoid spaces (ICS).
* Presence of Subfoveal neuroretinal detachment (SND) and height of serous macular detachment.
* The presence and size, and localization of hyperreflective foci (HF) within the retina.
* The disorganisation of the inner retinal layers (DRIL).
* The presence of vitreomacular traction.
* The integrity of the outer retinal layers, (ellipsoid zone (EZ) and external limiting membrane (ELM)).

E. Theinjectionprocedure:

The surgical notes will be reviewed from the patient's files to report the injection procedure, preparations and complications.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with centre-involving DME (CI-DME) who are treatment-naïve.
* Central macular thickness (CMT) of 300 microns or more will be accepted as DME.

Exclusion Criteria:

* Media opacities affecting OCT imaging (corneal pathologies, dense cataracts, vitreous opacities, etc).
* Patients with any other retinal vascular diseases (retinal vein occlusion, central serrous chorioretinopathy, age-related macular degeneration, etc).
* Patients who have had previous intravitreal injections or Laser treatment.
* Patients who underwent previous vitreoretinal surgeries.
* Patients with recent history of undergoing cataract surgery.
* Patients with uncontrolled glaucoma or ocular inflammations (eg: vitritis).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diabetic macular Oedema patients who are treatment naïve.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2026-01-16 (Estimated); Study Completion 2026-01-16 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | one month
  Visual acuity assessment pre and post injection will be recorded
Central subfield thickness | one month
  Central subfield thickness assessment pre and post injection will be recorded
Intraretinal cystoid spaces | one month
  Intraretinal cystoid space location, size and bridging will be recorded pre and post injection
Subfoveal neuroretinal detatchment | one month
  Presence and extent of Subfoveal neuroretinal detatchment assessed pre and post injection will be recorded
Hyperreflective foci | one month
  number and locatio of Hyperreflective foci assessed pre and post injection will be recorded
Outer retinal layer integrity | one month
  Outer retinal layer integrity assessment pre and post injection will be recorded
Disorganised inner retinal layers | one month
  Disorganised inner retinal layers assessment pre and post injection will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt